CLINICAL TRIAL: NCT06340269
Title: Feasibility Pilot Study to Evaluate the Safety and Performance of the MEX-CD1 Medical Device in Acute on Chronic Liver Failure (ACLF)
Brief Title: Feasibility Pilot Study to Evaluate the Safety and Performance of the MEX-CD1 Medical Device in ACLF
Acronym: MexACLF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mexbrain (Industry)
Collaborators: Slb Pharma (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PJ2308-0025
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Acute on Chronic Liver Failure; Multiple Organ Failure
Keywords: ACLF; Intensive Care Unit; Iron; Hemodialysis
MeSH Terms: conditions — Acute-On-Chronic Liver Failure; Multiple Organ Failure

STUDY DESIGN:
Intervention Model Description: Prospective, national, monocentric, single-arm, open label, feasibility pilot clinical trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MEX-CD1 Slow Low volume CVVHD (Experimental): Patients enrolled in the treatment arm will receive 3 sessions of MEX-CD1 treatment in addition to standard of care
  Interventions: Device: MEX-CD1 Dialysis

INTERVENTIONS:
Device: MEX-CD1 Dialysis — MEX-CD1 is a hyper-chelating colloidal solution that can be added to the dialysate to be used in Slow low-volume continuous veno-venous hemodialysis. One treatment will last 3 hours and 20 minutes.
  Patients enrolled are hospitalized in Intensive Care Unit.
  Other Names: Slow Low-volume continuous veno-venous haemodialysis

SUMMARY:
The goal of this clinical trial is to test the MEX-CD1 hemodialysis medical device in patients suffering from ACLF. The main questions it aims to answer are:

* Is the device safe when used according to the instructions for use?
* Does the device work as expected by removing the excess of free iron from the blood?

Patients will receive 3 MEX-CD1 Slow Low volume CVVHD within 1 week.

DETAILED DESCRIPTION:
This study investigates the safety and performance of the MEX-CD1 slow low volume CVVHD device in patients suffering from ACLF.

Acute-on-chronic liver failure (ACLF) is defined as a syndrome in patients with acutely decompensated cirrhosis, associated with single or multiple organ failures, and characterized by a high short-term mortality. ACLF is frequently triggered by a precipitating event (alcoholic hepatitis, infection, gastrointestinal haemorrhage) and characterized by an intense systemic inflammatory response driven per pathogen-associated molecular patterns (PAMPs) and/or damage-associated molecular patterns (DAMPs) responsible of the development of organs failure through tissues hypoperfusion, immune-mediated tissue damages and mitochondrial dysfunction.

Very importantly, ACLF is a very dynamic syndrome that has potential for reversibility. It is hypothesized that the extraction of non-transferrin bound iron (NTBI) could break down the vicious cycle of the excessive inflammatory responses, reduce oxidative stress and inhibit pathogen proliferation in ACLF patients.

As a consequence, it is hypothesized that the extraction of NTBI could promote improvement of ACLF grade n to ACLF grade n-1 or no ACLF. It is hypothesized that the extraction of NTBI could stop the progression of ACLF by preventing further organ failures and by reducing bacterial infection. Thereby, the extraction of NTBI could restore the eligibility of ACLF patients to liver transplantation, and, with or without liver transplantation, allow an earlier discharge from intensive care and prolong survival.

The proposed medical device, by combining dialysis to a hyper-chelating colloidal dialysate (MEX-CD1), specifically extracts free iron from the blood.

All patients enrolled in this study will receive 3 MEX-CD1 Slow Low volume CVVHD within 1 week. The duration of each MEX-CD1 Slow Low volume CVVHD session is 3h20.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects ≥18 years and ≤80 years
* Subject is able to provide informed consent to participate in the study, otherwise written consent must be obtained on behalf of the subject by a next of kin or legal representative in accordance with local ethical and legal requirements
* History of an acute decompensation event (including but not limited to ascites, gastrointestinal bleeding, hepatic encephalopathy and/or acute bacterial infections), occurring within ≤6 weeks of screening
* Cirrhosis (diagnosed based on clinical, biological, morphological parameters or liver biopsy)
* Subject with:

  * ACLF Grade 2, 3a or 3b based on the CLIF-C OF score
  * Under continuous renal replacement therapy (CRRT) or any organ support device that requires catheter placement

Exclusion Criteria:

* Subjects with acute or sub-acute liver failure without an underlying cirrhosis
* Subjects not considered appropriate for full active treatment including organ support or those with a Do Not Attempt Cardio-Pulmonary Resuscitation order (DNACPR)
* Subjects who have received any investigational drug or device within 30 days of dosing or who are scheduled to receive another investigational drug or device in the course of the study; concomitant observational studies are allowed
* Evidence of uncontrolled seizures
* In females: known pregnancy or lactating
* Patients with a known allergy to shellfish
* Patients for who, in the opinion of the investigator, it would be unsafe to be considered for the study
* Vulnerable population according to Articles 64 to 68 of the Regulations (EU) 2017/745 on Medical Devices
* Patient with weight < 30 kg

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-06-21 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
SADE for Safety purpose | From the enrollment until the last visit, assessed up to 7 days.
  The safety will be assessed by percentage of subjects who discontinued MexACLF due to a serious adverse device event (SADE) between Day 1 and Day 7.

SECONDARY OUTCOMES:
SAE for Safety purpose | From the start of the first MEX-CD1 treatment until the last visit, assessed up to 7 days.
  The safety will be assessed by the percentage of patients who experience at least one related Serious Adverse Event (SAE) between Day 1 and Day 7.
Performance of MEX-CD1 | 3 hours and 20 minutes; from treatment start (0 hours) to treatment end (3h20)
  The performance of the MEX-CD1 slow low-volume CVVHD treatment in terms of iron extraction will be measured by the amount of iron extracted in the dialysate bags per treatment.
Change in Acute on Chronic Liver Failure (ACLF) Grade | Between the screening visit and the last visit, assessed up to 7 days.
  Assessment of the change in ACLF Grade between the baseline and the end of study Min value = 0 (no ACLF) Max value=3b (Worse outcome)
Change in CLIF-C ACLF score | Between the screening visit and the last visit, assessed up to 7 days.
  Assessment of the change in Chronic Liver Failure-Consortium (CLIF-C) ACLF score between the baseline and the end of study. CLIF-C ACLF = 10 × (0.33 × CLIF-C OFs + 0.04 x Age + 0.63 × ln (WBC count)-2)
  CLIF-OFs= Chronic Liver Failure Consortium Organe Failure Min value=6 (No organe Failure) Max value=18 (6 organe failures)
Improvement in individual organ function | Between the screening visit and the last visit, assessed up to 7 days.
  Assessment of the change in individual organ function by using the CLIF sequential OF score
  From 1 (no organe failure) to 3 (worse outcome) for the 6 organes below:
  Liver ; kidney ; Brain ; Coagulation ; Circulation ; Respiratory
Development of secondary infection | Between the screening visit and the last visit, assessed up to 7 days.
  Assessment of development of secondary infection by need for new antibiotic therapy
Status of ICU | Between the screening visit and the last visit, assessed up to 28 days.
  Length of stay in ICU
hospital discharge | Between the screening visit and the last visit, assessed up to 28 days.
  Length of stay at hospital
Mortality | Between the screening visit and the last visit, assessed up to 28 days.
  Assessment of the survival rate

CONTACTS AND LOCATIONS:
Overall Officials: Céline GUICHON, MD, Principal Investigator — Hôpital Croix Rousse, Service d'hépatologie et gastroentérologie
Locations (2):
- France (2):
  - Hôpital Croix Rousse, Service d'hépatologie et gastroentérologie, Lyon, Auvergne-Rhône-Alpes
  - CHU Pontchaillou, Rennes